CLINICAL TRIAL: NCT02073734
Title: Effects of Preoperative Dexamethasone on Postoperative Quality of Recovery Following Vaginal Reconstructive Surgery: A Randomized Controlled Trial
Brief Title: Effects of Preoperative Dexamethasone Study on QOL After Vaginal Reconstructive Surgery for POP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12136-12-081
Record Dates: First submitted 2013-04-25; First posted 2014-02-27 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Pelvic Organ Prolapse; PONV
Keywords: pelvic organ prolapse surgery; dexamethasone; postoperative nausea and vomiting; peroperative administration
MeSH Terms: conditions — Pelvic Organ Prolapse; Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Sterile normal saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8mg/IV
  Arms: Dexamethasone
Drug: Placebo — Placebo given IV
  Arms: Placebo

SUMMARY:
The investigators hypothesize that preoperative administration of 8 mg IV dexamethasone will benefit patients' perceived quality of recovery after surgery.

DETAILED DESCRIPTION:
This is a randomized controlled trial involving single administration of 8 mg Dexamethasone per IV preoperatively among women undergoing vaginal reconstructive surgery for pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-81 years old who are scheduled to undergo a major vaginal reconstructive surgery, including hysterectomy with or without hysterectomy

Exclusion Criteria:

* Daily use of steroids or antiemetic agents such as Zofran, Reglan, Compazine and Phenargan within one month of surgery
* Regional anesthesia for surgical procedure
* Chronic pain requiring opioid treatment daily
* History of allergy to the study medication
* Severe renal and liver disease
* Pregnancy
* Non English speaking
* Psychiatric disorder that will preclude completion of questionnaires
* Minor surgery that does not involve overnight admission
* Surgery that does not involve hysterectomy or vaginal intraperitoneal apical suspension
* Hypersensitivity reaction to steroids
* Evidence of systemic fungal infection
* Evidence of any systemic infection
* Uncontrolled diabetes

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be scores on the 40- item quality of recovery scoring system (QoR-40). | up to 20-24 hours after surgery
  The QoR-40 is a validated standardized questionnaire that assesses the dimensions of physical functioning, mental health, cognitive functioning, symptoms, role and social functioning, general health perceptions, sleep and energy

SECONDARY OUTCOMES:
To determine if dexamethasone has positive impact on other clinical recovery variables such as nausea, vomiting and pain. | 20-24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Pauls, MD, Study Director — TriHealth Good Samaritan Hospital; Rachel N Pauls, MD, Principal Investigator — TriHeath Good Samaritan Hospital
Locations (1):
- Triheath, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pauls RN, Crisp CC, Oakley SH, Westermann LB, Mazloomdoost D, Kleeman SD, Ghodsi V, Estanol MV. Effects of dexamethasone on quality of recovery following vaginal surgery: a randomized trial. Am J Obstet Gynecol. 2015 Nov;213(5):718.e1-7. doi: 10.1016/j.ajog.2015.05.061. Epub 2015 May 29. PMID 26032041